CLINICAL TRIAL: NCT00500994
Title: Neurobiological Studies of Functional Movement Disorders and Non-Epileptic Seizures
Brief Title: Neurobiology of Functional Movement Disorder and Non-Epileptic Seizures
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 070190; 07-N-0190
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Movement Disorders
Keywords: Conversion Disorder; Psychogenic Movement Disorders; Non-Epileptic Seizure; Functional Magnetic Resonance Imaging (fMRI); Genetic Polymorphisms
MeSH Terms: conditions — Movement Disorders; Conversion Disorder; Seizures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- fMRI study (Experimental): subjects receiving MRI
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — The imaging study will use a block design to (i) optimize amygdala activation to emotionally valenced images, (ii) to optimize analysis of PPI and (iii) to optimize the go/no-task design. G. T2-sensitive functional images will be obtained on a MRI system with a 1.5 Tesla superconducting magnet and a standard head coil. An echo planar image sequence (TR=2500msec, TE=33 msec, 90 flip angle) with 30 contiguous 2mm thick coronal oblique slices with 1 mm interslice gap centered over the amygdala, tilted 30 to the anterior, to improve susceptibility artifact. Three-dimensional anatomical images will be taken for the co-registration of the functional images.

SUMMARY:
This study is part of a series of studies that will explore how the mind and the brain work to cause episodes of uncontrollable shaking in people who have no known underlying brain or medical disorder. The study is conducted at NIH and at the Brown University Rhode Island Hospital.

Healthy volunteers and people with functional movement disorders (FMD) or non-epileptic seizures (NES) who are 18 years of age or older may be eligible for this study.

Patients with NES have 3 teaspoons of blood drawn. The blood is tested for two genes that are normally found in healthy individuals to see if they are found more frequently in patients with uncontrolled shaking.

Patients with FMD have blood drawn for testing and also undergo functional magnetic resonance imaging (fMRI) to look at how the brain functions while the subject performs a specific task. MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. During the scan, the subject lies on a table that can slide in and out of the scanner, a metal cylinder. The scan lasts about 60 to 90 minutes, during which the subject may be asked to lie still for up to 10 minutes at a time and to perform tasks, such as identifying the gender of faces shown on a screen.

Healthy volunteers may have blood drawn for genetic testing or fMRI or both.

DETAILED DESCRIPTION:
Objectives:

The study investigates the neurobiological correlates of conversion disorder (CD). The primary objectives are to investigate in CD patients:

* The role of emotional valence in an implicit emotional processing task (COMPLETE)
* The frequency of the 5HTTLPR S/S genotype
* Structural differences in grey matter of the brain as detected by voxel-based morphometry (VBM)
* The neural correlates of fear conditioning and fear extinction in a fear learning fMRI task
* The neural correlates of interoceptive activity in a Interoceptive Attention fMRI task
* Identifying the cortical physiology correlated with making a movement following a go command.
* Identifying the cortical physiology correlated with not making a movement following a no-go command.
* Identifying the cortical physiology correlated with planning to move or not move following a choose go-no go command.

Exploratory objectives are to investigate in CD patients:

* The frequency of several gene polymorphisms that are implicated in stress and affective disorder, including 5HTTLPR S/S (serotonin receptor), COMT (catechol-o-methyltransferase enzyme), Val/Met BDNF (brain-derived neurotrophic factor) and FKBP5 rs1360780 genotypes, as well as other polymorphisms or mutations to be determined later. Additionally, epigenetic data will be explored.
* The levels of salivary cortisol as a measure of stress.
* The heart rate variability, as a measure of autonomic nervous system function. (COMPLETE)
* Structural differences in white matter of the brain as detected by diffusion tensor imaging (DTI)
* The resting state BOLD fMRI signal
* The impact of the caregiver's attitude on the patients' symptoms
* The relationship between hemodynamic responses in regions implicated in interoception and self-reported measures of interoceptive attention, as well as behavioral and motor symptom severity

Study population:

We intend to study adult patients with diagnoses of functional movement disorders (FMD) seen by the Human Motor Control Section clinic (HMCS), patients with diagnoses of psychogenic non-epileptic seizures (PNES) seen by the Epilepsy clinic and healthy volunteers. Up to 12 healthy volunteers will be for the EEG-EMG sub-study. The PNES patient group will include patients seen at Rhode Island Hospital. Additionally, we would like to study caregivers of patient's with FMD who are enrolled un protocol 07-N-0190.

Design:

An assessment for psychiatric diagnoses and measurement scales will be administered to the FMD and PNES patients, healthy volunteer controls and caregivers.

* Functional MRI (fMRI): emotional processing will be studied using a gender identification task with differing emotional valences. (COMPLETE) Limbic processing will also be studied using a fear learning fMRI task. Resting state BOLD fMRI signal will also be obtained.
* Anatomical MRI: VBM and DTI will be performed using anatomical MRI sequences collected during the fMRI scanning or subsequent dedicated anatomical MRI sessions.
* Genetics: blood will be collected for testing.
* Stress biomarkers: saliva will be collected for testing. [EVALUATION IN HEALTHY VOLUNTEERS COMPLETE].
* Autonomic nervous system function: electrocardiogram (EKG) will be obtained to determine heart rate variability. [COMPLETE].
* Event related potentials: 64-channel EEG and surface EMG will be recorded during a go , no-go and choose go-no go behavioral task.
* EEG will be recorded during the resting state condition (five minutes with eyes open and five minutes with eyes closed).

Outcome measures:

* fMRI study: blood oxygenation level dependent (BOLD) signal in the regions of interest during a gender identification task (primary) [COMPLETE], in regions of interest during a fear learning task (primary), as well as resting state BOLD signal (exploratory). EEG resting state data will be compared and correlated with the fMRI resting state data.
* Anatomical MRI: VBM (primary) and DTI (exploratory)
* Genetics: (a) S/S genotype of the serotonin transporter promoter region polymorphism. (primary) (b) Polymorphism frequency of several genes related to affective disorders and/or stress (exploratory)
* Stress biomarkers: salivary cortisol levels (exploratory). [EVALUATION IN HEALTHY VOLUNTEERS COMPLETE]
* Autonomic nervous system function: heart rate variability as measured by EKG (exploratory). [COMPLETE]
* Psychological profile scales: scores exploratory.
* The relationship between hemodynamic responses in regions implicated in interoception and self-reported measures of IA, motor symptoms and behavioral ratings (exploratory)
* EEG-EMG study: Characteristics of event related cortical potentials correlated with simple behavioral motor tasks in healthy volunteers. Differences between go and no-go potentials will be identified and quantified. This analysis will allow planning a properly powered study for patients with functional movement disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:

General Inclusion Criteria for FMD patients:

* Diagnosis of clinically definite FMD utilizing Fahn and Williams criteria. The diagnosis must be made by a neurologist
* Able to give informed consent
* Age 18 or older

General Inclusion Criteria for Caregivers:

* Age 18 or older
* Able to give informed consent
* Takes care of a patient with FMD patient enrolled in protocol 07-N-0190 for 10 or more weekly hours.

General Inclusion Criteria for PNES patients:

* Diagnosis of PNES based on recording of patient s typical episode during 24 h video-EEG without concomitant EEG changes. The diagnosis must be made by a neurologist.
* Able to give informed consent
* Age 18 or older

General Inclusion Criteria for Healthy Volunteers:

* Able to give informed consent
* Age 18 or older

EXCLUSION CRITERIA:

General exclusion criteria for FMD patients:

* Significant neurological disorders (primary or comorbid) such as neurodegenerative disorders, stroke, movement disorders or epilepsy
* Inflammatory disorders or autoimmune disorders active within the last 6 months
* Patients with psychotic disorders or manic depression or active substance abuse within the last 6 months
* Current suicidal ideation
* Disease severity requiring inpatient treatment

Additional exclusion criteria for FMD patients for MRI:

* Patients with movement symptoms at rest that may substantially inhibit resolution, comfort, or safety of MRI
* Previous history of or MRI findings consistent with brain tumors, strokes, trauma or arterial venous malformations
* History of traumatic brain injury with loss of consciousness or amnesia lasting greater than a few seconds
* Contraindication to MRI
* Pregnancy
* Significant medical illness
* Patients with current post-traumatic stress disorder
* Patients on tricyclic antidepressants or antiepileptic medications 2 weeks prior to testing

General exclusion criteria for PNES patients:

* Significant neurological disorders (primary or comorbid) such as neurodegenerative disorders, stroke, movement disorders or epilepsy
* Inflammatory disorders or autoimmune disorders active within the last 6 months
* Patients with psychotic disorders or active substance abuse within the last 6 months
* Current suicidal ideation
* Disease severity requiring inpatient treatment

General exclusion criteria for healthy volunteers:

* Significant neurological disorders (primary or comorbid) such as neurodegenerative disorders, stroke, movement disorders or epilepsy
* History of DSM IV-defined schizophrenia, schizoaffective disorder, bipolar disorder or major depression with psychosis
* History of psychotic disorders or manic depression or active substance abuse within the last 6 months
* Subjects with post-traumatic stress disorder
* Subjects on antidepressants or antiepileptic medications
* Inflammatory disorders or autoimmune disorders active within the last 6 months

Additional exclusion criteria for healthy volunteers for MRI:

* Previous history of or MRI findings consistent with brain tumors, strokes, trauma or arterial venous malformations
* Contraindication to MRI
* Pregnancy
* Significant medical illness

General Exclusion Criteria for Caregivers:

* History of DSM-IV defined Schizophrenia, Schizoaffective Disorder, Bipolar Disorder, Major depression with psychotic features (by interview).
* Active substance abuse within the past 6 months (by interview).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2007-10-05 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
fMRI study: blood oxygenation level dependent (BOLD) signal in the regions of interest during a gender identification task | throughout
  fMRI BOLD signal change focusing on regions of interest during emotional valence task
Genetics: S/S genotype of the serotonin transporter promoter region polymorphism. | throughout
  The S/S genotype of the 5HTTLPR polymorphism
Anatomical MRI: VBM | throughout
  Structural grey matter brain data

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Joo Cho, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Rhode Island Hospital (RIH), Providence, Rhode Island

REFERENCES:
- [Derived] Waugh RE, Parker JA, Hallett M, Horovitz SG. Classification of Functional Movement Disorders with Resting-State Functional Magnetic Resonance Imaging. Brain Connect. 2023 Feb;13(1):4-14. doi: 10.1089/brain.2022.0001. Epub 2022 Jun 16. PMID 35570651
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-N-0190.html